CLINICAL TRIAL: NCT02188563
Title: Efficacy and Impact of a Comprehensive Smoking Cessation Intervention During Radiation for Upper Aerodigestive Cancers
Brief Title: A Comprehensive Smoking Cessation Intervention Duration Radiation for Upper Aerodigestive Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1407; NA_00089912 (Other: JHM IRB); P50DE019032 (NIH)
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2015-05

CONDITIONS: Tobacco Use Disorder; Head and Neck Neoplasms; Thoracic Neoplasms; Radiation
Keywords: Smoking cessation; Head and neck neoplasms; Lung neoplasms; Thoracic neoplasms; Radiation
MeSH Terms: conditions — Tobacco Use Disorder; Head and Neck Neoplasms; Thoracic Neoplasms; Smoking Cessation; Lung Neoplasms

ARMS (2):
- Comprehensive intervention (Experimental): New evidence-based comprehensive smoking cessation intervention including several elements that have proven successful in non-cancer patients but not used for cancer patients before.
  Interventions: Other: Comprehensive smoking cessation intervention
- Enhanced usual care (Active Comparator): Intervention consistent with the U.S. Department of Health and Human Services guidelines for tobacco treatment.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Other: Comprehensive smoking cessation intervention
  Arms: Comprehensive intervention
Behavioral: Enhanced usual care
  Arms: Enhanced usual care

SUMMARY:
Smoking is the greatest risk factor for upper aerodigestive cancers (thoracic or head and neck) and negatively impacts survival and other outcomes, but many patients have difficulty quitting after their diagnosis. Smoking cessation interventions for cancer patients thus far have had limited success. This is a pilot randomized controlled trial designed to determine if a new comprehensive, evidence-based smoking cessation intervention can improve quit rates for cancer patients who smoke.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of head and neck or thoracic (including lung) cancer
* Undergoing radiation at Johns Hopkins Radiation Oncology for 5 or more weeks
* English-speaking and able to provide informed consent
* Smoked any cigarettes in previous 14 days

Exclusion Criteria:

* Palliative radiation
* Undergoing stereotactic radiosurgery
* Pregnant or breastfeeding

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 8 weeks
  Smoking cessation will be defined as BOTH (1) self-reported 7-day abstinence from smoking and (2) exhaled carbon monoxide level of 8 or lower as biochemical confirmation of abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Gypsyamber D'Souza, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health, Department of Epidemiology
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440